CLINICAL TRIAL: NCT03685968
Title: A Comparison of the King Vision® Channeled, King Vision® Non-Channeled, and Glidescope® Video Intubation Systems in Patients at Risk for Difficult Intubation - A Pilot Study
Brief Title: King Vision® and GlideScope® in Difficult Airways
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: King Systems Corporation (Industry)
Responsible Party: Principal Investigator, Carin A. Hagberg, Chief Academic Officer and Division Head of Anesthesiology, Critical Care, and Pain Medicine, M.D. Anderson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-13-0024
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Airway Management

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Glidescope AVL (Experimental)
  Interventions: Device: Video laryngoscopes
- King Vision Channeled VL (Experimental)
  Interventions: Device: Video laryngoscopes
- King Vision Non-Channeled (Standard) VL (Experimental)
  Interventions: Device: Video laryngoscopes

INTERVENTIONS:
Device: Video laryngoscopes — Patients were randomized into one of the three groups through a computer generated randomization schedule. Patients in group A (N= 75) will be intubated using the GlideScope® AVL, patients in group B (N= 75) will be intubated using the King Vision Channeled VL; patients in group C (N=75) will be intubated using the King Vision Video Laryngoscope with Standard (non-channeled) Blade. Patients will only be tested with one device. All patients will be intubated using a conventional ETT.

SUMMARY:
There are several advantages of video laryngoscopy; especially their ability to provide superior glottis visualization, as compared to traditional laryngoscopy.1-3 The purpose of this three arm study was to compare the safety and efficacy of the King Vision® Video Intubation Systems (AMBU-King Systems, Denmark) to the Cobalt GlideScope® (Verathon Medical Inc., USA) in patients with anticipated difficult airways.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Mallampati III-IV
* Neck circumference > 43cm
* Reduced mouth opening (< 4cm) or 3 Finger breath's (patient's own)
* Thyromental distance < 6cm

Exclusion Criteria:

* Mallampati I-II
* Neck circumference < 43cm
* Documented 'easy' intubation
* Previous history of failed intubation and failed bag-mask ventilation
* Under 18 years of age
* ASA IV
* Known unstable cervical spine injury
* Presentation for an emergency surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2013-03-06 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carin A Hagberg, MD, Study Chair — M.D. Anderson Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hagberg CA, Iannucci D, Goodrich A. A comparison of the glottic view obtained with the Macintosh Video Laryngoscope in anesthetized, paralyzed, apneic patients. Direct view vs video monitor. Anesthesiology 2003; 103: A1501.
- [Background] Hagberg C, Matuszczak M, Ellis S, et al. A randomized comparison of laryngoscopy techniques using the video laryngoscope and the traditional Macintosh laryngoscope in obese patients. Anesthesiology 2005; 103: A1420.
- [Background] Hagberg C, Vogt-Harenkamp C, Bogomolny Y, et al. A comparison of laryngoscopy techniques using the video laryngoscope and the traditional Macintosh laryngoscope in potentially difficult to intubate patients. Anesth Analg 2005; 100: S-212.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from the adult surgical operating rooms of 2 academic hospitals, Lyndon Baines Johnson General Hospital and Memorial Hermann Hospital - Texas Medical Center, in Houston, TX from August 2013 to December 2015.
Groups:
- Glidescope AVL: Group A: Patients were randomized into one of the three groups through a computer-generated randomization schedule. Patients in group A (N= 75) were intubated utilizing the GlideScope® AVL.
- King Vision Channeled VL: Group B: Patients were randomized into one of the three groups through a computer-generated randomization schedule. Patients in group B (N= 75) were intubated utilizing the King Vision Channeled VL.
- King Vision Non-Channeled (Standard) VL: Group C: Patients were randomized into one of the three groups through a computer-generated randomization schedule. Patients in group C (N=75) were intubated utilizing the King Vision Video Laryngoscope with Standard (Non-Channeled) Blade.
Period: Overall Study
Arm/Group | Glidescope AVL | King Vision Channeled VL | King Vision Non-Channeled (Standard) VL
Started | 75 | 75 | 75
Completed | 75 | 75 | 75
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glidescope AVL | King Vision Channeled VL | King Vision Non-Channeled (Standard) VL | Total
Number analyzed (Participants) | 75 | 75 | 75 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 68 | 63 | 65 | 196
  >=65 years | 7 | 12 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (11.8) | 48.0 (15.2) | 50.0 (14.2) | 48.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 41 | 40 | 120
  Male | 36 | 34 | 35 | 105
Height (in) [Mean (Standard Deviation); unit: inches] | 66.7 (4.2) | 66.4 (4.3) | 66.4 (4.2) | 66.5 (4.2)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 117.5 (20.3) | 116.2 (25.5) | 116.8 (21.5) | 116.8 (22.4)
BMI (kg/m2) [Mean (Standard Deviation); unit: kilogram per meter square] | 41.2 (8.1) | 41.4 (9.9) | 41.1 (8.5) | 41.2 (8.8)
Neck Circumference (cm) [Mean (Standard Deviation); unit: centimeters] | 47.1 (4.3) | 47.1 (4.7) | 47.9 (4.3) | 47.3 (4.4)
Interincisor distance (cm) [Mean (Standard Deviation); unit: centimeters] | 4.1 (1.0) | 4.1 (0.9) | 4.1 (1.0) | 4.1 (0.9)
Thyromental distance (cm) [Mean (Standard Deviation); unit: centimeters] | 6.8 (1.7) | 6.8 (1.9) | 7.1 (1.7) | 6.9 (1.7)
Sternomental distance (cm) [Mean (Standard Deviation); unit: centimeters] | 13.4 (2.3) | 13.6 (2.3) | 13.7 (2.1) | 13.5 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Overall Successful Tracheal Intubation for All 3 Video Laryngoscopes - GSAVL, KVChVL and KVNChVL
Description: The overall intubation success rates for all 3 video laryngoscopes - GSAVL, KVChVL and KVNChVL
Time Frame: During laryngoscopy and endotracheal tube placement
Measure: Count of Participants; unit: Participants
Arm/Group | Glidescope AVL | King Vision Channeled VL | King Vision Non-Channeled (Standard) VL
Number analyzed (Participants) | 75 | 75 | 75
Participants | 72 | 61 | 72

2. Secondary Outcome: First-attempt Successful Intubation for All 3 Video Laryngoscopes - GSAVL, KVChVL and KVNChVL
Description: The overall first-attempt success rates for all 3 video laryngoscopes - GSAVL, KVChVL and KVNChVL
Time Frame: During laryngoscopy and endotracheal tube placement
Measure: Count of Participants; unit: Participants
Arm/Group | Glidescope AVL | King Vision Channeled VL | King Vision Non-Channeled (Standard) VL
Number analyzed (Participants) | 75 | 75 | 75
Participants | 64 | 53 | 67

3. Other Pre Specified Outcome: Final Intubation Time for All 3 Video Laryngoscopes - GSAVL, KVChVL and KVNChVL
Description: Total time for placing the endotracheal tube (ETT) through the vocal cords
Time Frame: During laryngoscopy and endotracheal tube placement
Population: Group A: 3 participants excluded due to protocol deviations. Group B: 8 participants excluded due to protocol deviations, 2 participant had failed intubation, 4 participants had device failure.
  Group C: 2 participants excluded due to protocol deviations, 1 participant had device failure.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Glidescope AVL | King Vision Channeled VL | King Vision Non-Channeled (Standard) VL
Number analyzed (Participants) | 72 | 61 | 72
seconds | 46.1 (27.4) | 44.9 (21.5) | 47.0 (24.3)

ADVERSE EVENTS:
Time Frame: Postoperatively in the PACU
Description: (Other Adverse Events) Group A: 3 participants excluded due to protocol deviations, 8 participants lost to follow up.
  Group B: 8 participants excluded due to protocol deviations, 2 participant lost to follow up.
  Group C: 2 participants excluded due to protocol deviations, 3 participant lost to follow up.
Arm/Group | Glidescope AVL | King Vision Channeled VL | King Vision Non-Channeled (Standard) VL
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 26/64 | 23/65 | 22/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Glidescope AVL (N=64) | King Vision Channeled VL (N=65) | King Vision Non-Channeled (Standard) VL (N=70)
Hoarseness (General disorders) | 26 | 23 | 22 — Hoarseness in voice postoperatively
Sore Mouth (General disorders) | 9 | 5 | 7 — Sore Mouth postoperatively
Sore neck (General disorders) | 9 | 4 | 7 — Sore neck postoperatively
Sore jaw (General disorders) | 4 | 1 | 2 — Sore jaw postoperatively
Dysphonia (General disorders) | 7 | 3 | 5 — Dysphonia postoperatively
Dysphagia (General disorders) | 13 | 14 | 9 — Dysphagia postoperatively
Alteration of tongue (General disorders) | 2 | 0 | 2 — Alteration of tongue postoperatively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No